CLINICAL TRIAL: NCT03775707
Title: Lenvatinib Plus Programmed Cell Death Protein-1 (PD-1) Antibody for Intermediate-stage Hepatocellular Carcinoma Beyond Up-to-seven Criteria
Brief Title: Lenvatinib Plus PD-1 Antibody for Intermediate-stage HCC Beyond Up-to-seven Criteria
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol modification
Sponsor: Shi Ming (Other)
Responsible Party: Sponsor-Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S063
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2018-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Lenvatinib; PD-1 Antibody; BCLC B stage; Beyond up-to-seven criteria
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib Plus PD-1 (Experimental): Participants received lenvatinib capsules 12 milligram (mg) based on the participant's body weight greater than or equal to (>=) 60 kilogram (kg) or 8 mg based on the participant's body weight less than (<) 60 kg at baseline, orally, once daily (QD) in continuous 14-day treatment cycles, and received 3mg/kg PD-1 antibody intravenously every 2 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Drug: Lenvatinib; Drug: PD-1 antibody

INTERVENTIONS:
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.
Drug: PD-1 antibody — 3mg/kg intravenously every 2 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of lenvatinib combined with PD-1 antibody for patients with intermediate-stage hepatocellular carcinoma (HCC) beyond up-to-seven criteria

DETAILED DESCRIPTION:
Lenvatinib was non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma, and PD-1 antibody was effective and tolerable in patients with advanced hepatocellular carcinoma. No study has evaluated the efficacy and safety of lenvatinib plus PD-1 antibody. Thus, the investigators carried out this prospective study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage B
* Beyond up-to-seven criteria (hepatocellular carcinomas with seven as the sum of the size of the largest tumor [in cm] and the number of tumors)
* Eastern Cooperative Oncology Group performance status of 0 to 1
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not applicable for transarterial chemoembolization, surgical resection, and local ablative therapy.
* The following laboratory parameters:

Platelet count ≥ 75,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 30 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3 Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 12 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.

SECONDARY OUTCOMES:
progression free survival (PFS) | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on mRECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions.
Adverse Events | 12 months
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China